CLINICAL TRIAL: NCT05682664
Title: Luchtbrug Junior: Online Monitoring for Young Children With Preschool Wheeze
Brief Title: Luchtbrug Junior: the Next Step
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Luchtbrug Junior
Record Dates: First submitted 2022-12-19; First posted 2023-01-12 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: eHealth; Telemedicine; Wheezing
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Usual care for children with preschool wheeze consist of regular visits to the outpatient clinic every three months after starting the study, while in between these visits contact with the healthcare team is by telephone as needed. At inclusion and at every outpatient clinical visits (e.g. 3, 6, 9 and 12 months), parents/caregivers will be asked to update the healthcare team on disease symptoms by completing a digital version of Test for Respiratory and Asthma Control in Kids (TRACK) questionnaire.
  Interventions: Other: Usual care
- Luchtbrug Junior (intervention) (Experimental): Online monitoring via Luchtbrug Junior will replace 50% of the outpatient visits. Children in the intervention group will be monitored online monthly by a digital version of TRACK.
  Interventions: Other: Luchtbrug Junior (online monitoring)

INTERVENTIONS:
Other: Luchtbrug Junior (online monitoring) — Online monitoring via Luchtbrug Junior will replace 50% of the outpatient visits. Children in the intervention group will be monitored online monthly by a digital version of TRACK.
  Arms: Luchtbrug Junior (intervention)
Other: Usual care — Routine outpatient clinical visits every 3 months.
  Arms: Usual care

SUMMARY:
Rationale:

The introduction of e-health in the monitoring and management of patients with chronic conditions can be beneficial and efficient. The introduction of an online monitoring and management tool, "Luchtbrug", for children 6-16 yrs of age with asthma while reducing 50% of visits to the outpatient clinic, results in similar or improved asthma control while reducing costs. It is highly likely that this concept of e-health is suitable for other chronic conditions. Therefore the aim of the study is to investigate the added value of online monitoring and management of children with preschool wheeze (2-6 yrs of age).

Objective: To assess whether the number of symptom free days can be improved using online monitoring and disease management via Luchtbrug Junior, while reducing the number of outpatient clinic visits by 50%

Study design: Prospective multicentre (n=6) randomised trial in which disease management via Luchtbrug Junior will be compared with usual care.

Follow-up: 12 months.

Study population: children aged 2-6 yrs with preschool wheezing (multiple episode of cough, wheeze and dyspnoea).

Intervention (if applicable): Children will be randomised into usual care (n=135) or partly online care via Luchtbrug Junior (n = 135)

Main study parameters/endpoints:

Primary objective: Number of symptom free days (SFDs) based on the TRACK questionnaire, during the last four weeks of the study (measured at 12 months).

Secondary objectives:

Healthcare consumption: unscheduled visits Emergency Department (ED) or outpatient clinic, unscheduled phone calls, hospital admissions) Questionnaires into: Quality of Life (QoL), cost-effectiveness (direct and indirect costs), self-management of patients, adherence to treatment, satisfaction of parents/caregivers.

Usual care consists of regular visits to the outpatient clinic every 3 months after starting the study. In between visits contact with the healthcare team is by telephone as needed. At 3, 6, 9 and 12 months, patients will be asked to complete the TRACK questionnaire.

Online care using Luchtbrug Junior will include visits to the outpatient clinic every 6 months after starting the study. In between visits, parents/caregivers of the patient will be asked to answer the digital version of TRACK questionnaire monthly, therefore the parents/caregivers will received email-reminders. Appropriate feedback on their TRACK-scores will be provided by their healthcare team within two working days. Any interventions such as adjustment of treatment are at the judgment of the treating pediatrician. Therapy adherence will be monitored during the study by using smart inhalers.

DETAILED DESCRIPTION:
Introduction of online monitoring and disease management The introduction of e-health in the monitoring and management of patients with chronic conditions can be beneficial and efficient for patients and/or their parents/caregivers, healthcare professionals, the healthcare system and society in general. This option has become even more attractive during the global pandemic but is likely to remain an innovation that will last. Furthermore, when e-health can (partly) replace usual care (visits to the outpatient clinic), this is likely to reduce the financial burden of healthcare/society and introduction of e-health for chronic conditions while reducing visits to the outpatient clinic fits well with the transition project of the Dutch Ministry of Health, "de juiste zorg op de juiste plek", the right kind of care on the right location.

Previously, in a multicentre randomized trial in 8 Dutch hospitals it has been demonstrated that the introduction of an online monitoring and management tool, using online eHealth platform "Luchtbrug", for children 6-16 years with asthma, can reduce the amount of outpatient visits needed by 50% while maintaining the same level of asthma control and reducing healthcare costs. Subsequently, this platform was further implemented and investigated in 14 hospitals to identify the barriers and facilitators for successful implementation as well as studying the experiences and perceptions of our patients and healthcare professionals on using the platform. Luchtbrug is now used in the daily patient care for over 500 children with asthma in more than 20 Dutch hospitals and its costs are now reimbursed with support of Dutch Health Insurance companies and the Dutch Healthcare Authority.

Online management of children with preschool wheeze Almost 60% of children younger than six years old experience multiple episodes with cough, wheeze and dyspnea without any serious underlying condition. The majority don't require any medical treatment and improve spontaneously with age. However, in about 5% of the Dutch children aged 2-5 years (n ≈ 45.000) symptoms are more severe and require regular medical care, unscheduled health visits and/or hospital admissions.

Traditional medical care for these children consists of three to six scheduled outpatient clinic visits per year, during which pediatricians monitor treatment response and adjust the treatments accordingly. For many pediatric departments this is a considerable volume of patients, constituting a significant impact not only on patients and their caretakers, but also on the medical capacity of these hospitals.

Nevertheless, this implies that the patient is 'out of sight' for the remaining 350 days per year. With the introduction of e-Health with remote monitoring, patients can be managed much more closely while also reducing the amount of traditional consultations.

It is highly likely that Luchtbrug is also suitable for managing children with preschool wheeze (2-6 years old). However, in contrast to older children, the concept of online monitoring in preschool wheezing has barely been studied or evaluated in large randomized controlled trials. Therefore the aim of the study is to develop and study an eHealth platform for children with preschool wheeze called Luchtbrug Junior.

Luchtbrug Junior

Luchtbrug Junior is a web-based and smartphone (app) application. It is only accessible for parents/caregivers of registered children with preschool wheeze and their healthcare team (specialized nurse and paediatrician). It can be regarded as an extension of the regular outpatient clinic and has several modules:

1. An information module, with frequently asked questions, background information about disease symptoms and demonstrative movies
2. A secure and private section including:

   1. A monitoring section to enable frequent monitoring of symptoms through respiratory questionnaires once every month
   2. An individual and personalised treatment plan, including rescue plan
   3. A communication section in which parents/caregivers can communicate easily, freely and safely 24/7 with their healthcare team with guaranteed feedback within two working days.
   4. An overview to monitor treatment adherence and abnormal use of rescue medication by using smartinhalers.

In this proposed multicentre randomized controlled trial, the aim is to answer the following research question using Luchtbrug Junior: can the number of symptom free days be improved using online monitoring and disease management in children with preschool wheeze while reducing the number of outpatient clinic visits by 50%?

ELIGIBILITY:
Inclusion criteria

* Children aged 2 to 6 years with a doctor's diagnosis of preschool wheeze
* Children have an indication for regular follow-up of at least one year by a paediatrician because of respiratory symptoms;
* Children are treated with inhaler medication, including inhaled corticosteroids;
* A history of three episodes of wheezing managed by a healthcare professional of which at least one was observed by a paediatrician in the last 12 months prior to the study, or:
* At least one hospital admissions due to pulmonary symptoms before inclusion.
* Informed consent of parents/caregivers

Exclusion criteria

* Underlying chronic cardiopulmonary or neuromuscular condition, or known recurrent aspirations;
* Underlying syndromes associated with pulmonary comorbidities;
* Prematurity <36 weeks after gestation;
* Inability of parents/caregivers/caretakers to understand and/or read Dutch;
* No access to a smartphone and/or internet.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change of Symptom free days / TRACK | TRACK questionnaire at baseline, 3, 6 , 9 and 12 months
  Number of symptom free days (SFDs) based on the TRACK questionnaire during the last four weeks of the study (measured at 12 months). The amount of SFDs varies from 0 days to 30 days a month. A higher number indicates more symptom free days in the last four weeks of the study

SECONDARY OUTCOMES:
Healthcare consumption | Through study completion (follow-up of 12 months)
  Healthcare consumption:
  * Number of unscheduled emergency department (ED) visits,
  * Number of unscheduled outpatient clinic visits,
  * Number of unscheduled phone calls,
  * Number of hospital admissions, and
  * Amount of medication prescriptions of systemic corticosteroids.
Paediatric caregivers quality of life (PACQLQ) (by Juniper) | Both groups will complete the PACQLQ at baseline, and 6 and 12 months
  This questionaire focuses in how parents/caregivers are limited in their own quality of life due to the child's disease. The questionnaire with a 1 week recall period consists of 13 items in two domains: emotional functioning and activity. Each items is scored using a 7-point scale, with 7 being indicative for optimal asthma related QoL. Items were all equally weighted and the overall PACQLQ score was measured by the mean of these item-scores. Minimal important difference for clinical relevance is 0.7 points
Self-management of parents/caregivers | At baseline and at 6 and 12 months
  The degree of self management will be assessed by a self-made questionnaire containing open questions and will be used for qualitative analyses. After completing the questionnaire, 10-15 parents/caregivers will be interviewed to obtain. The aim is to assess more detailed information about these self management skills and any change thereof during the study.
Cost-effectiveness | At baseline and every 3 months for 1 year
  Cost-effectiveness: medical/direct costs and social/indirect costs by completing a cost diary
Patient Reported Experiences Measures (PREMs) | At baseline, after 6 and 12 months.
  Self-made qualitative questionnaires will be used to assess PREMs: patients/caregivers experiences, satisfaction, concerns, needs and thoughts about eHealth. When more detailed information is needed based on thisx questionnaire, a random sample of participants will be interviewed.
Therapy adherence | At baseline and every 3 months for a year by completing TAI12. In the intervention group continuously monitoring by using smart inhalers
  Adherence to therapy measured by TAI12 and continuously in the intervention group by using smart inhalers. TAI12 is the Test of the Adherence of Inhalers. In this questionnaire, 10-items are completed by participants, each item scored from 1 to 5 (where 1 was the worst possible score and 5 was the best possible score), with a range from 10 to 50. The other two items are assessed by the health care professional and scored as 1 or 2 (where 1 was bad and 2 was good), with a range from 2 to 4. An erratic and deliberate non-adherent behavioral pattern was defined in the presence of scores ≤24 for items #1 to #5 and items #6 to #10, respectively. The unwitting pattern was defined in the presence of a score 1 in at least one of the #11 or #12 items of the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lara van den Wijngaart, MD, PhD, Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: No